CLINICAL TRIAL: NCT06138327
Title: A Phase 1b, Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, 2-Period Crossover Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of an Oral Administration of BMN 255 in Participants With Non-Alcoholic Fatty Liver Disease (NAFLD) And Hyperoxaluria
Brief Title: A Study of BMN 255 in Participants With Non-Alcoholic Fatty Liver Disease And Hyperoxaluria
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was withdrawn because BioMarin decided to end the overall development program. The study withdrawal was not due to any patient safety concerns.
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 255-102
Record Dates: First submitted 2023-10-18; First posted 2023-11-18 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Hyperoxaluria; Nonalcoholic Fatty Liver Disease; Kidney Stone
Keywords: Kidney Stones; Nonalcoholic Fatty Liver Disease; Hyperoxaluria; NAFLD; MASLD; Metabolic Dysfunction-associated Steatotic Liver Disease
MeSH Terms: conditions — Hyperoxaluria; Non-alcoholic Fatty Liver Disease; Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMN 255 Investigational drug arm (Experimental): Oral administration of BMN 255 at a dose of 100mg per day for 7 days in Treatment Period 1 or 2
  Interventions: Drug: BMN 255
- Placebo Comparative drug arm (Placebo Comparator): Oral administration of Placebo at a dose of 100mg per day for 7 days in Treatment Period 1 or 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMN 255 — Oral Capsule
  Arms: BMN 255 Investigational drug arm
Drug: Placebo — Oral Capsule
  Arms: Placebo Comparative drug arm

SUMMARY:
The purpose of this study is to test the safety of BMN 255 and to learn about the effect BMN 255 has on you and your hyperoxaluria associated with NAFLD, and compare these effects with a placebo.

The primary safety objective of the study is to assess the safety and tolerability of daily oral doses of BMN 255 in adult participants with NAFLD and hyperoxaluria.

The primary efficacy objective of the study is to assess 24-hour urine oxalate levels (24-hour urine collection corrected for BSA) following daily oral doses of BMN 255 in adult participants with NAFLD and hyperoxaluria.

ELIGIBILITY:
Inclusion Criteria:

1. History of NAFLD with a liver fat content ≥ 8.0%, as determined by Fibroscan (transient elastography) or magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) during screening.
2. Hyperoxaluria, as defined by 24-hour urine oxalate excretion ≥ 45 mg/24 hours/1.73m2 at 2 independent assessments during screening. The pre-dose 24-hour urine oxalate measure at Day 1 will be used for baseline but will not be required for inclusion in the study
3. History of kidney stones (at least 1 stone prior to screening based on medical history); participants with a known personal or family history of cystinuria or cystine kidney stones, calcium phosphate stones, struvite stones, or urate stones should not be included.
4. Contraceptive use by men and women use throughout the study period
5. Participants must be capable of giving signed informed consent

Exclusion Criteria:

1. Clinical history (including family history) or genetic analyses consistent with primary hyperoxaluria (Type 1, 2, or 3).
2. History or current evidence of inflammatory bowel disease (including, but not limited to: Crohn's disease, ulcerative colitis, celiac disease / gluten-sensitive enteropathy) or evidence of chronic fat malabsorption (steatorrhea) due to any cause (eg, pancreatic insufficiency).
3. Significant history or clinical manifestation of any other allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator. Participants with Type II diabetes will be permitted to enroll but must meet the concomitant therapy requirements listed below.
4. Use or intend to use any prescription medications/products within 14 days prior to Period 1 check-in, other than permitted oral medications to treat controlled hypertension, dyslipidemia and/or to lower triglycerides, and oral anti-hyperglycemic agents (AHAs), including, but not limited to, metformin, sulfonylureas, and dipeptidyl peptidase IV (DPP-IV) inhibitors, if approved by the investigator. Participants who require insulin injections, glucagon-like peptide-1 agonists, pioglitazone, or vitamin E ≥ 800 mg should not be included in the study.

   Note: Participants receiving lipid-modifying therapies and participants with controlled hypertension and/or diabetes must have been on a stable treatment regimen (medication, dose strength, dose interval) for 12 weeks prior to screening and no change in that regimen should be anticipated for the entire duration of this study (ie, from screening to final follow-up visit).
5. Confirmed diagnosis or NASH or evidence of hepatic cirrhosis, based on clinical assessment (eg, physical examination), historical liver biopsy or other prior imaging study, or a liver stiffness value ≥ 14 kPa during the FibroScan® examination at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint is the incidence of adverse events in adult participants with NAFLD and hyperoxaluria | Treatment Periods 1 & 2 through a 15 day follow-up after period 2. Each treatment period is 7 days separated by a 7-9 day washout period.
  - Including but not limited to acute liver or kidney injury

SECONDARY OUTCOMES:
To characterize the daily oral dose plasma pharmacokinetics of BMN 255 in adult participants with NAFLD and hyperoxaluria. | Day 1, Day 7 of treatment periods 1 & 2, each treatment period is 7 days separated by a 7-9 day washout period and Day 15
  Area under the plasma concentration-time curve (AUC)
To characterize the daily oral dose plasma pharmacokinetics of BMN 255 in adult participants with NAFLD and hyperoxaluria. | Day 1, Day 7 of treatment periods 1 & 2, each treatment period is 7 days separated by a 7-9 day washout period and Day 15
  Maximum observed concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (7):
- United States (7):
  - University of Alabama - Department of Urology, Birmingham, Alabama
  - ProSciento, Inc., Chula Vista, California
  - ProSciento, Inc., Chula Vista Isles, Florida
  - Georgia Clinical Research, LLC, Lawrenceville, Georgia
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - Centricity Research, Columbus, Ohio
  - Prolato Clinical Research Center, Houston, Texas